CLINICAL TRIAL: NCT05165121
Title: Comparison of Hearing Aid Fitting Outcomes Between Self-fit and Professional Fit for MDHearing Smart Hearing Aids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MDHearingAid (Industry)
Collaborators: Central Michigan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1001
Record Dates: First submitted 2021-11-23; First posted 2021-12-21 (Actual); Results first posted 2023-07-06 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2021-12

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Human Factors (Other): The purpose of the human factor study was to verify the feasibility of self-fitting MDHearing Smart hearing aid by listeners with a mild to moderate sensorineural hearing loss.
  Interventions: Device: MDHearing smart hearing aid
- Clinical Study (Other): The clinical study included two groups of subjects (self-fit and professional-fit groups) with the main purpose to compare the fitting outcomes between the two fitting groups. The professional-fit group aimed to show whether the MDHearing Smart hearing aids can be fitted by audiology professional on each user reliably and if each user can benefit from using the MDHearing smart hearing aids. The self fit group intended to show whether the MDHearing Smart hearing aids can be fitted by each user reliably and if each user can use the MDHearing app on their smartphone or tablet to make adjustments to achieve a good aided benefit.
  Interventions: Device: MDHearing smart hearing aid

INTERVENTIONS:
Device: MDHearing smart hearing aid — air conduction hearing aid with app support

SUMMARY:
Hearing aids are commonly used to help people with hearing loss hear better in daily listening environments. MDHearing Smart hearing aids are designed to use the MDHearing app to adjust hearing aids to each individual's hearing loss. This study intends to show whether the MDHearing Smart hearing aids can be fitted by each user reliably and if each user can use the MDHearing app on their smartphone or tablet to make adjustments to achieve good aided benefit, which will be compared to those fitted by audiology professionals. This study includes three components: human factor study, self-fit study, and professional-fit study. The information obtained will be useful for both audiology professionals and people with impaired hearing.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old
* At least one air conduction threshold above 15dB HL.
* All air conduction thresholds must be under 60dB HL

Exclusion Criteria:

* Signs of outer or middle ear pathology
* Greater than 60db HL hearing loss at any frequency.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2020-09-21 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-09-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yunfang Zheng, Sc.D. CCC-A, Principal Investigator — Central Michigan University
Locations (1):
- Central Michigan University, Mount Pleasant, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Clinical Study - Self Fit Group: The clinical study included two groups of subjects (self-fit and professional-fit groups) with the main purpose to compare the fitting outcomes between the two fitting groups. The self fit group intended to show whether the MDHearing Smart hearing aids can be fitted by each user reliably and if each user can use the MDHearing app on their smartphone or tablet to make adjustments to achieve a good aided benefit.
  MDHearing smart hearing aid: air conduction hearing aid with app support
- Clinical Study - Professional Fit Group: The clinical study included two groups of subjects (self-fit and professional-fit groups) with the main purpose to compare the fitting outcomes between the two fitting groups. The professional-fit group aimed to show whether the MDHearing Smart hearing aids can be fitted by audiology professional on each user reliably and if each user can benefit from using the MDHearing smart hearing aids.
  MDHearing smart hearing aid: air conduction hearing aid with app support
Period: Overall Study
Arm/Group | Human Factors | Clinical Study - Self Fit Group | Clinical Study - Professional Fit Group
Started | 20 | 36 | 35
Completed | 20 | 32 | 32
Not Completed | 0 | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Human Factors | Clinical Study - Self Fit Group | Clinical Study - Professional Fit Group | Total
Number analyzed (Participants) | 20 | 36 | 35 | 91
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 15 | 20 | 20 | 55
  >=65 years | 5 | 16 | 15 | 36
Age, Continuous [Mean (Full Range); unit: years] | 52 [19 to 74] | 62 [31 to 76] | 58 [31 to 79] | 52 [19 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 18 | 21 | 49
  Male | 10 | 18 | 14 | 42
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20 | 36 | 35 | 91

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Improvement at 1 Month as Measured by the Abbreviated Profile of Hearing Aid Benefit (APHAB) and Speech Spatial Qualities 12 (SSQ 12) Scale.
Description: Comparison of aided benefit between the self-fit group and the professional fit group as measured by the Abbreviated Profile of Hearing Aid Benefit (APHAB) and Speech Spatial Qualities 12 (SSQ 12). The lowest possible score on the APHAB is 1% with the highest score being 99%. A higher score indicates improvement. On the SSQ, the scores range from 0 to 10 with a higher score indicating hearing perfectly in that situation. For the SSQ Part B, the scores range from -5 to +5 with a higher score indicating improved hearing for that situation.
Time Frame: 1 month
Measure: Count of Participants; unit: Participants
Groups:
- APHAB - Self Fit Group; APHAB - Professional Fit Group: Comparison of aided benefit between the self-fit group and the professional fit group as measured by the Abbreviated Profile of Hearing Aid Benefit (APHAB). The lowest possible score on the APHAB is 1% with the highest score being 99%. A higher score indicates improvement
- SSQ 12 - Self Fit Group; SSQ 12 - Professional Fit Group: Comparison of aided benefit between the self-fit group and the professional fit group as measured by the Speech Spatial Qualities 12 (SSQ 12). On the SSQ, the scores range from 0 to 10 with a higher score indicating hearing perfectly in that situation.
- SSQ 12 Part B - Self Fit Group; SSQ 12 Part B - Professional Fit Group: Comparison of aided benefit between the self-fit group and the professional fit group as measured by the Speech Spatial Qualities 12 (SSQ 12). For the SSQ Part B, the scores range from -5 to +5 with a higher score indicating improved hearing for that situation.
Arm/Group | APHAB - Self Fit Group | APHAB - Professional Fit Group | SSQ 12 - Self Fit Group | SSQ 12 - Professional Fit Group | SSQ 12 Part B - Self Fit Group | SSQ 12 Part B - Professional Fit Group
Number analyzed (Participants) | 32 | 32 | 32 | 32 | 32 | 32
Participants | 32 | 32 | 32 | 32 | 32 | 32

2. Primary Outcome: Human Factors Study: Percentage of Participants Able to Use Hearing Aids Both With and Without Guidance.
Description: Subjects are able to use the hearing aids while using the app and manuals as guidance. Ease of use will be self reported by the subjects as to whether the task was able to be completed without guidance, able to be completed with guidance from the manual, or unable to be completed. Participants self-reported their comfort level with hearing aids and with technology in general. Participants sat with a researcher to note if tasks were able to be completed without guidance, with guidance from the manual, or unable to be completed.
  This group was separate from the Self Fit group and the Professional Group.
Time Frame: 1 hour
Measure: Number; unit: percentage of participants
Groups:
- Usability of the Hearing Aids: Subjects had to complete the following tasks:
  Unbox the hearing aids. Download the MDHearing Smart app to a personal smartphone. Register for the app. Place a battery in the hearing aids. Use the app to pair the hearing aids to the smartphone via Bluetooth. Use the app to take the personalization profile. Use the app to adjust the volume, program, noise reduction, microphone direction, bass, treble, and mid pitched settings.
  Turn off the hearing aids.
Arm/Group | Usability of the Hearing Aids
Number analyzed (Participants) | 20
percentage of participants | 100

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the time of the study. One hour for the Human Factors portion of the study and thirty days for the Clinical Trials portion of the study.
Groups:
- Clinical Study - Self-fit Group: The clinical study included two groups of subjects (self-fit and professional-fit groups) with the main purpose to compare the fitting outcomes between the two fitting groups. The self fit group intended to show whether the MDHearing Smart hearing aids can be fitted by each user reliably and if each user can use the MDHearing app on their smartphone or tablet to make adjustments to achieve a good aided benefit.
  MDHearing smart hearing aid: air conduction hearing aid with app support
- Clinical Study - Professional-fit Group: The clinical study included two groups of subjects (self-fit and professional-fit groups) with the main purpose to compare the fitting outcomes between the two fitting groups. The professional-fit group aimed to show whether the MDHearing Smart hearing aids can be fitted by audiology professional on each user reliably and if each user can benefit from using the MDHearing smart hearing aids.
  MDHearing smart hearing aid: air conduction hearing aid with app support
Arm/Group | Human Factors | Clinical Study - Self-fit Group | Clinical Study - Professional-fit Group
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/36 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/36 | 0/35
Other Adverse Events (participants affected / at risk) | 0/20 | 0/36 | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-07-13): https://cdn.clinicaltrials.gov/large-docs/21/NCT05165121/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-21): https://cdn.clinicaltrials.gov/large-docs/21/NCT05165121/SAP_001.pdf